CLINICAL TRIAL: NCT00224575
Title: Therapeutical Impact of a Reassessment Strategy in the Diagnosis of Coronary Heart Disease in Elderly
Brief Title: Reassessment Strategy in the Diagnosis of Coronary Heart Disease in Elderly
Acronym: IRIDIA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of recruitment period
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOM03099
Record Dates: First submitted 2005-09-13; First posted 2005-09-23 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Myocardial Ischemia
Keywords: Veterans
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Diagnosis strategy and subsequent therapeutic reassessment All patients are in that arms. They all receive the diagnosis reassessment strategy.
  Interventions: Other: diagnosis reassessment; Other: Diagnosis strategy and subsequent therapeutic reassessment

INTERVENTIONS:
Other: diagnosis reassessment — Strategy of diagnosis reassessment following a decision tree.
  Other Names: no other names to specified
Other: Diagnosis strategy and subsequent therapeutic reassessment — Performed by geriatricians, following a decision tree, based on medical history, electrocardiogram, cardiac echotomography and stress scintigraphy

SUMMARY:
Despite the effectiveness of beta-blockers and antiplatelet agents for secondary prevention of coronary heart disease, this treatments are underused in the elderly because of diagnosis uncertainty and underuse of efficient treatment.

in a first time, diagnosis reassessment with invasive technique if necessary. in a second time, treatment reassessment.

DETAILED DESCRIPTION:
not desired

ELIGIBILITY:
Inclusion Criteria:

* patients 75 of age or older hospitalized in a geriatric service and suspect of coronary heart disease

Exclusion Criteria:

* acute myocardial infarction

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 260 (Actual)
Dates: Start 2004-11; Primary Completion 2005-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
therapeutical impact of a reassessment strategy in the diagnosis of coronary heart disease in elderly | during hospitalization

SECONDARY OUTCOMES:
part link, in the treatment modification, with diagnosis reassessment and the part link with treatment optimization, death and rehospitalization in the subsequent 6 and 12 months | during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: legrain sylvie, Principal Investigator — APHP
Locations (1):
- Hopital Bichat, Paris, Paris, France